CLINICAL TRIAL: NCT00530946
Title: A Multi-Center, Randomized Study To Evaluate Efficacy And Safety Of A Fixed Combination Therapy Of Amlodipine And Atorvastatin In The Treatment Of Concurrent Hypertension And Hyper-LDL-Cholesterolemia
Brief Title: A Randomized Study To Evaluate Efficacy And Safety Of A Fixed Combination Therapy Of Amlodipine And Atorvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3841058
Record Dates: First submitted 2007-09-13; First posted 2007-09-18 (Estimated); Results first posted 2009-04-13 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Hypercholesterolemia
MeSH Terms: conditions — Hypertension; Hypercholesterolemia | interventions — Amlodipine; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CI-1038 2.5mg/5mg (Active Comparator)
  Interventions: Drug: Amlodipine 2.5mg/Atorvastatin 5mg
- CI-1038 2.5mg/10mg (Active Comparator)
  Interventions: Drug: Amlodipine 2.5mg/Atorvastatin 10mg
- CI-1038 5mg/5mg (Active Comparator)
  Interventions: Drug: Amlodipine 5mg/Atorvastatin 5mg
- CI-1038 5mg/10mg (Active Comparator)
  Interventions: Drug: Amlodipine 5mg/Atorvastatin 10mg

INTERVENTIONS:
Drug: Amlodipine 2.5mg/Atorvastatin 5mg — Single pill combination, dosed once daily for 8 weeks
  Arms: CI-1038 2.5mg/5mg
Drug: Amlodipine 2.5mg/Atorvastatin 10mg — Single pill combination, dosed once daily for 8 weeks
  Arms: CI-1038 2.5mg/10mg
Drug: Amlodipine 5mg/Atorvastatin 5mg — Single pill combination, dosed once daily for 8 weeks
  Arms: CI-1038 5mg/5mg
Drug: Amlodipine 5mg/Atorvastatin 10mg — Single pill combination, dosed once daily for 8 weeks
  Arms: CI-1038 5mg/10mg

SUMMARY:
To assess the changes in the trough Systolic Blood Pressure (SBP) and the percent changes in Low Density Lipoprotein-Cholesterol (LDL-C) from baseline at Week 8 in the treatment period

ELIGIBILITY:
Inclusion Criteria:

* The out-patient with concurrent hypertension and hyper-LDL-cholesterolemia is a male or female >=20 to <80 years of age at Visit 1.
* The SBP at Visit 4 (Week -1) and Visit 5 (Week 0) is continuously SBP >=140 mmHg and <180 mmHg,
* LDL-C >=140 mg/dL and <250 mg/dL at Visit 3 (Week -2) and 4 (Week -1).

Exclusion Criteria:

* Subjects who had experienced the following coronary artery disease within the past 3 months.
* Myocardial infarction
* Receiving PCI（percutaneous coronary intervention）or CABG (coronary artery bypass grafting)
* Any clinically meaningful valvular disease
* Subjects with a history of cerebrovascular diseases such as stroke or transient ischemic attack within the past 3 months.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Japan (17):
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu-shi, Fukuoka
  - Pfizer Investigational Site, Kurume-shi, Fukuoka
  - Pfizer Investigational Site, Maebaru-shi, Fukuoka
  - Pfizer Investigational Site, Annaka, Gunma
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Teine, Hokkaido
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Yamashitachō, Naka-ku, Kanagawa-ken
  - Pfizer Investigational Site, Kita-ku, Osaka
  - Pfizer Investigational Site, Koshigaya-shi, Saitama
  - Pfizer Investigational Site, Chōfu, Tokyo
  - Pfizer Investigational Site, Kiyose, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shinagawa-Ku, Tokyo
  - Pfizer Investigational Site, Shinagawa, Tokyo
  - Pfizer Investigational Site, Osaka

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841058&StudyName=A%20Randomized%20Study%20To%20Evaluate%20Efficacy%20And%20Safety%20Of%20A%20Fixed%20Combination%20Therapy%20Of%20Amlodipine%20And%20Atorvastatin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty (20) centers in Japan
Pre-assignment Details: A total of 301 subjects entered the 6-week diet observation period and the end of diet observation period, 165 subjects who met all the inclusion criteria for the treatment period and had no conflict to exclusion criteria were randomized to 4 CI-1038 groups.
Groups:
- CI-1038 2.5 mg/5 mg: Amlodipine 2.5 mg/Atorvastatin 5 mg single pill combination (CI-1038 2.5mg/5mg)
- CI-1038 2.5 mg/10 mg: Amlodipine 2.5 mg/Atorvastatin 10 mg single pill combination (CI-1038 2.5 mg/10 mg)
- CI-1038 5 mg/5 mg: Amlodipine 5 mg/Atorvastatin 5 mg single pill combination (CI-1038 5 mg/5 mg)
- CI-1038 5 mg/10 mg: Amlodipine 5 mg/Atorvastatin 10 mg single pill combination (CI-1038 5 mg/10 mg)
Period: Overall Study
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Started | 43 | 41 | 41 | 40
Completed | 41 | 39 | 40 | 38
Not Completed | 2 | 2 | 1 | 2
Not completed — Adverse Event | 1 | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Noncompliance | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg | Total
Number analyzed (Participants) | 43 | 41 | 41 | 40 | 165
Age, Customized [Number; unit: participants]
  <20 years | 0 | 0 | 0 | 0 | 0
  20 to 44 years | 8 | 3 | 4 | 5 | 20
  45 to 64 years | 20 | 21 | 23 | 23 | 87
  >=65 years | 15 | 17 | 14 | 12 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 25 | 22 | 98
  Male | 20 | 13 | 16 | 18 | 67
Region of Enrollment [Number; unit: participants]
  Japan | 43 | 41 | 41 | 40 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Description: Value at Week 8 minus value at baseline
Time Frame: 8 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
mm Hg | -16.6 (1.65) | -15.9 (1.69) | -21.8 (1.69) | -18.9 (1.71)

2. Primary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol
Description: Percent of "value at Week 8 minus value at baseline" over value at baseline
Time Frame: 8 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
Percent Change | -37.2 (1.49) | -42.5 (1.52) | -34.3 (1.52) | -40.6 (1.54)

3. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Each Observation Point
Description: Value at Week 2, Week 4, or Week 8 minus value at baseline
Time Frame: 2 weeks, 4 weeks, and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
mm Hg
  Week 2 | -12.8 (9.63) | -13.5 (10.18) | -19.2 (10.53) | -16.0 (9.01)
  Week 4 | -14.2 (10.26) | -14.6 (12.33) | -20.2 (11.08) | -19.6 (11.03)
  Week 8 | -16.8 (11.40) | -15.3 (11.59) | -21.3 (10.07) | -18.7 (11.24)

4. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Each Observation Point
Description: Value at Week 2, Week 4, or Week 8 minus value at baseline
Time Frame: 2 weeks, 4 weeks , and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
mm Hg
  Week 2 | -4.9 (6.23) | -6.0 (6.05) | -8.1 (6.24) | -8.2 (6.38)
  Week 4 | -5.3 (4.96) | -8.2 (7.13) | -9.4 (6.19) | -9.2 (6.62)
  Week 8 | -7.7 (6.34) | -8.7 (8.06) | -12.0 (6.31) | -9.9 (6.57)

5. Secondary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol From Baseline to Each Observation Point
Description: Percent of "value at Week 2, Week 4, or Week 8 minus value at baseline" over value at baseline
Time Frame: 2 weeks, 4 weeks , and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
Percent Change
  Week 2 | -34.8 (9.11) | -42.5 (11.00) | -32.8 (9.15) | -40.2 (13.52)
  Week 4 | -37.4 (7.67) | -43.8 (9.30) | -35.0 (9.19) | -41.8 (9.53)
  Week 8 | -37.6 (7.80) | -42.9 (10.28) | -34.2 (9.22) | -40.8 (11.28)

6. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Each Observation Point
Description: Percent of "value at Week 2, Week 4, or Week 8 minus value at baseline" over value at baseline
Time Frame: 2 weeks, 4 weeks , and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
Percent Change
  Week 2 | -24.2 (6.86) | -30.5 (8.44) | -23.0 (7.22) | -28.3 (10.04)
  Week 4 | -26.6 (6.36) | -31.5 (7.08) | -24.7 (7.64) | -28.6 (7.44)
  Week 8 | -26.1 (6.01) | -30.0 (8.43) | -23.4 (7.78) | -28.2 (8.73)

7. Secondary Outcome: Percent Change in High Density Lipoprotein-Cholesterol From Baseline to Each Observation Point
Description: Percent of "value at Week 2, Week 4, or Week 8 minus value at baseline" over value at baseline
Time Frame: 2 weeks, 4 weeks , and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
Percent Change
  Week 2 | 7.7 (12.11) | 8.3 (10.70) | 6.6 (9.12) | 9.9 (10.32)
  Week 4 | 7.2 (8.16) | 7.9 (13.03) | 9.3 (13.24) | 11.9 (13.28)
  Week 8 | 7.2 (10.86) | 7.5 (13.27) | 9.7 (10.59) | 10.8 (9.66)

8. Secondary Outcome: Percent Change in Triglycerides From Baseline to Each Observation Point
Description: Percent of "value at Week 2, Week 4, or Week 8 minus value at baseline" over value at baseline
Time Frame: 2 weeks, 4 weeks , and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
Percent Change
  Week 2 | -15.1 (33.82) | -27.4 (22.48) | -16.2 (20.00) | -23.9 (24.51)
  Week 4 | -14.2 (25.31) | -25.7 (18.15) | -15.1 (22.42) | -23.2 (28.55)
  Week 8 | -14.1 (19.72) | -21.1 (21.68) | -10.8 (31.42) | -24.0 (25.15)

9. Secondary Outcome: Change in Low Density Lipoprotein-Cholesterol/ High Density Lipoprotein-Cholesterol Ratio (LDL-C/HDL-C) From Baseline to Each Observation Point
Description: Value at Week 2, Week 4, or Week 8 minus value at baseline
Time Frame: 2 weeks, 4 weeks, and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
Ratio
  Week 2 | -1.2 (0.58) | -1.4 (0.42) | -1.1 (0.49) | -1.3 (0.53)
  Week 4 | -1.3 (0.41) | -1.4 (0.42) | -1.2 (0.56) | -1.4 (0.49)
  Week 8 | -1.2 (0.37) | -1.4 (0.44) | -1.2 (0.52) | -1.4 (0.52)

10. Secondary Outcome: Change in Total Cholesterol/ High Density Lipoprotein-Cholesterol Ratio (TC/HDL-C) From Baseline to Each Observation Point
Description: Value at Week 2, Week 4, or Week 8 minus value at baseline
Time Frame: 2 weeks, 4 weeks , and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
Ratio
  Week 2 | -1.3 (0.71) | -1.6 (0.49) | -1.2 (0.61) | -1.5 (0.64)
  Week 4 | -1.4 (0.48) | -1.6 (0.49) | -1.4 (0.69) | -1.6 (0.59)
  Week 8 | -1.3 (0.43) | -1.5 (0.51) | -1.4 (0.65) | -1.5 (0.62)

11. Secondary Outcome: Change in Apolipoprotein B From Baseline to Each Observation Point
Description: Value at Week 2, Week 4, or Week 8 minus value at baseline
Time Frame: 2 weeks, 4 weeks, and 8 weeks
Population: Full Analysis Set, Observed Cases
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Number analyzed (Participants) | 43 | 41 | 41 | 40
mg/dL
  Week 2 | -36.6 (12.55) | -45.8 (12.11) | -33.5 (9.86) | -44.4 (15.46)
  Week 4 | -40.1 (10.94) | -47.2 (10.20) | -36.6 (11.36) | -45.8 (13.79)
  Week 8 | -40.2 (9.65) | -46.4 (10.87) | -36.6 (12.27) | -45.1 (14.39)

ADVERSE EVENTS:
Arm/Group | CI-1038 2.5 mg/5 mg | CI-1038 2.5 mg/10 mg | CI-1038 5 mg/5 mg | CI-1038 5 mg/10 mg
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 6/43 | 7/41 | 8/41 | 8/40
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CI-1038 2.5 mg/5 mg (N=43) | CI-1038 2.5 mg/10 mg (N=41) | CI-1038 5 mg/5 mg (N=41) | CI-1038 5 mg/10 mg (N=40)
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 6 | 3 | 5 | 7
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.